CLINICAL TRIAL: NCT01341873
Title: Nursing Intervention for Family Caregivers of HCT Patients
Brief Title: Nursing Intervention in Supporting Family Caregivers of Patients Undergoing Stem Cell Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol was not funded by the NCI
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10235; NCI-2011-00574 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-21; First posted 2011-04-26 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Anxiety Disorder; Depression; Fatigue
MeSH Terms: conditions — Anxiety Disorders; Depression; Fatigue | interventions — Early Intervention, Educational; Methods; Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (FCI) (Experimental): FCs receive 4 sessions of an APN FCI beginning during the admission for transplant and continuing for up to 100 days after transplant.
  Interventions: Other: educational intervention; Other: psychosocial support for caregiver; Procedure: quality-of-life assessment; Other: questionnaire administration
- Group II (control) (Other): FCs receive standard supportive care.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Undergo APN FCI
  Other Names: intervention, educational
  Arms: Group I (FCI)
Other: psychosocial support for caregiver — Undergo APN FCI
  Arms: Group I (FCI)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies nursing intervention in supporting family caregivers (FCs) of patients undergoing stem cell transplant. A nursing intervention may help prepare FCs support the recovery of the patients

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the effects of an advanced practice nursing (APN) intervention for family caregivers (FCs) of hematopoietic cell transplant (HCT) patients in the experimental group on FC quality of life, psychological distress, caregiver burden, caregiver skills preparedness as compared to FCs in the control group.

II. Describe self-care behaviors for FCs of HCT patients and compare them between the experimental and control groups.

III. Describe resource use by FCs comparing the experimental and control groups.

IV. Identify subgroups of FCs who benefit most from the family caregiver intervention (FCI) in relation to sociodemographic characteristics, caregiver health status, and patient characteristics.

SECONDARY OBJECTIVES:

I. Describe family caregivers' satisfaction with the FCI.

OUTLINE: FCs are randomized to 1 of 2 groups.

GROUP I: FCs receive 4 sessions of an APN FCI beginning during the admission for transplant and continuing for up to 100 days after transplant.

GROUP II: FCs receive standard supportive care.

After completion of study, FCs are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The primary family caregiver as identified by a hematologic cancer patient who is scheduled for a single allogeneic bone marrow or stem cell transplant; the definition of a family caregiver for the purposes of this proposal refers to either a family member or friend that is identified by the patient as being the primary caregiver
* Living within a 50 mile radius of City of Hope

Exclusion Criteria:

* Caregivers who are unable to read English or Spanish consent forms
* Caregivers who live more than 50 miles from City of Hope

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Test the effects of an advanced practice nursing (APN) intervention for family caregivers (FCs) in the experimental group using questionnaires measuring quality of life and psychological distress as compared to the FCs in the control group. | 12 months after discharge
Test the effects of an advanced practice nursing (APN) intervention for family caregivers (FCs) in the experimental group using questionnaires measuring caregiver burden and skills preparedness as compared to the FCs in the control group. | 12 months after discharge
Through the use of questionnaires, comparison of self-care behaviors for FCs of Hematopoietic Cell Transplant (HCT) patients between the experimental and control groups | 12 months after discharge
Through the use of questionnaires, comparison of resource use between the experimental and control groups | 12 months after discharge
Through the use of questionnaires, identification of subgroups of FCs who benefit most from the Family Care Intervention (FCI) in relation to sociodemographic characteristics, caregiver health status, and patient characteristics | 12 months after discharge

SECONDARY OUTCOMES:
Through the use of questionnaires, measure FCs satisfaction with the FCI | 12 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSC, Principal Investigator — City of Hope Medical Center